CLINICAL TRIAL: NCT04660994
Title: Contribution of an Educational Game for Continuous Positive Pressure/Non-invasive Ventilation Therapeutic Education in Children
Acronym: YAPOUNI
Status: Withdrawn | Type: Observational
Why Stopped: Abandoned project
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200959; 2020-A01737-32 (Other: ID RCB number)
Record Dates: First submitted 2020-11-19; First posted 2020-12-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2022-12

CONDITIONS: Sleep Disordered Breathing
Keywords: Nocturnal continuous positive airway pressure therapy; Nocturnal non-invasive ventilation therapy; Sleep disordered breathing; Therapeutic education; Educational game; Therapeutic compliance; Motivation
MeSH Terms: conditions — Sleep Apnea Syndromes; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Therapeutic education: Children with disordered breathing requiring CPAP or NIV and followed-up by the pediatric non-invasive ventilation and sleep unit of Necker-Enfants Malades hospital.
- Therapeutic education and Yapouni educational game: Children with disordered breathing requiring CPAP or NIV and followed-up by the pediatric non-invasive ventilation and sleep unit of Necker-Enfants Malades hospital.
  Interventions: Other: Educational game

INTERVENTIONS:
Other: Educational game — The Yapouni educational game is based on a hot air balloon that will fly according to the number of hours the child has slept with his/her CPAP / NIV. Thus, the longer the child sleeps with his/her CPAP / NIV, the farther and higher his/her hot air balloon will fly in the sky. The game includes wild cards and rewards that are worked out with the child and his/her parents for an optimal individualized adaptation.
  The game is explained at Necker Hospital during the therapy education for CPAP/NIV and used at home for 1 month.
  Other Names: YAPOUNI
  Groups: Therapeutic education and Yapouni educational game

SUMMARY:
A growing number of children with obstructive sleep apnea syndrome (OSAS) or nocturnal alveolar hypoventilation syndrome are treated with continuous positive airway pressure (CPAP) or nocturnal non-invasive ventilation (NIV) therapy.

The compliance of the child and his caregivers with CPAP / NIV therapy may be challenging.

The use of an educational game (Yapouni) aims at improving communication around CPAP / NIV between the child and his caregivers, and may facilitate the compliance with CPAP / NIV at home, by increasing the motivation for using CPAP / NIV at home.

The aim of the study is to assess the parents' feelings regarding the use of CPAP / NIV on day 0 (D0) and one month (D30) later in a standard group: therapeutic education (TEP) versus a group: TEP + Yapouni.

DETAILED DESCRIPTION:
The study concerns children with severe obstructive sleep apnea syndrome and / or alveolar hypoventilation requiring the initiation of CPAP/NIV. Most of these children have associated diseases (craniofacial malformations, trisomy 21, Prader Willi syndrome or neuromuscular diseases) which are accompanied by an abnormality of nocturnal breathing causing abnormalities in gas exchange and abnormalities of architecture and quality of sleep, with deleterious consequences on neurocognitive, cardiovascular and metabolic functions. In the absence of other treatments, the initiation of CPAP or NIV during sleep can correct the respiratory anomalies and the deleterious consequences. Optimal compliance with treatment is therefore essential for its efficacy and therapeutic education (TEP) plays a key role.

The compliance of the child and his caregivers with CPAP / NIV therapy may be challenging.

The use of an educational game (Yapouni) aims at improving communication around CPAP / NIV between the child and his caregivers, and may facilitate the compliance with CPAP / NIV at home, by increasing the motivation for using CPAP / NIV at home.

The Yapouni educational game is based on a hot air balloon that will fly according to the number of hours the child has slept with his/her CPAP / NIV. Thus, the longer the child sleeps with his/her CPAP / NIV, the farther and higher his/her hot air balloon will fly in the sky. The game includes wild cards and rewards that are worked out with the child and his/her parents for an optimal individualized adaptation.

The aim of the study is to assess the parents' feelings regarding the use of CPAP / NIV on D0 and D30 later in a standard group: therapeutic education (TEP) versus a group: TEP + Yapouni.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 16 years old with severe obstructive sleep apnea syndrome and / or alveolar hypoventilation requiring the initiation of a treatment with CPAP / NIV in the pediatric non-invasive ventilation and sleep unit of Necker-Enfants Malades hospital.
* Child's caregivers not opposing to the patient's participation in research.

Exclusion Criteria:

* Non-communicating child.
* Child with major cognitive impairment.
* Child / parents not speaking French.
* Child in an unstable clinical condition.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 3 to 16 years old with severe obstructive sleep apnea syndrome and / or alveolar hypoventilation requiring the initiation of a treatment with CPAP / NIV in the pediatric non-invasive ventilation and sleep unit of Necker-Enfants Malades hospital.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Parents'feelings | Scale change from day 0 to day 30
  Quantitative score at the parental feelings questionnaire about the CPAP/NIV initiation process.
  Home made questionnaire of 5 questions with responses by visual analogue scale from 0 to 100; 0 is the worst feeling and 100 the best.

SECONDARY OUTCOMES:
Feeling of children | Scale change from day 0 to day 30
  Quantitative score of the questionnaire of feelings of the children about the CPAP/NIV initiation process.
  Home made questionnaire of 5 questions with responses by visual analogue scale from 0 to 10; 0 is the worst feeling and 10 the best.
Parents' concerns or difficulties | Scale change from day 0 to day 30
  Score on the parental concerns and difficulties questionnaire regarding the health of their children.
  Questionnaire of 6 questions of 7-level ordinal scale of answer; 0 is the worst feeling and 100 the best.
Family impact | Change from day 0 to day 30
  Pediatric Quality of Life Inventory, Parent-Proxy Report (PEDSQL) questionnaire on family impact of the child's illness (s) rated from 0 to 100, high results being associated with a better quality of life.
Functioning of the child | Change from day 0 to day 30
  Pediatric Quality of Life Inventory, Child-Self Report (PEDSQ) questionnaire on the child functioning rated from 0 to 100, high results being associated with a better quality of life.
Therapeutic compliance in hours | Change from day 8 to day 30
  Average number of hours of CPAP / NIV use per night.
Therapeutic compliance in days | Change from day 8 to day 30
  Average number of days of CPAP / NIV use.
Motivation of parents | Change from day 0 to day 30
  Parent motivation scale (adaptation of the situational motivation scale). Questionnaire of 9 questions of 7-level ordinal scale of answer ; 0 is the worst feeling and 100 the best.
Motivation of children | Change from day 0 to day 30
  Child motivation scale (adaptation of the situational motivation scale). Questionnaire of 3 questions with responses by visual analogue scale from 0 to 10; 0 is the worst score and 10 the highest motivation.
Parents competence | Change from day 0 to day 30
  Parents competence scale (adaptation of the perceived competence scale). Questionnaire of 4 questions of 5-level ordinal scale of answer; 0 is the worst feeling and 100 the best.
Children competence | Change from day 0 to day 30
  Children competence scale (adaptation of the perceived competence scale). Questionnaire of 2 questions with responses by visual analogue scale from 0 to 10; 0 is the worst score and 10 the highest competence feeling.
Effect of the TEP session on healthcare professionals | Change from day 0 to day 30
  Score at the questionnaire on the effect of the session on healthcare professionals.
  Questionnaire of 5 questions of 7-level ordinal scale of answer, the higher the score, the more positive the feeling ; 0 is the worst feeling and 100 the best.
Number of calls from parents | Day 30
  Number of calls from parents regarding to CPAP / NIV and Yapouni game.
Score on Yapouni questionnaire for parents | Change from day 8 to day 30
  Parents' evaluation of the game. Questionnaire of 5 questions of 7-level ordinal scale of answer, the higher the score, the more positive the appreciation ; 0 is the worst feeling and 100 the best.
Score on Yapouni questionnaire for children | Change from day 8 to day 30
  Evaluation of the game by children. Questionnaire of 3 questions with responses by visual analogue scale from 0 to 10; 0 is the worst score and 10 the highest appreciation.
Score on Yapouni questionnaire for healthcare professionals | Change from day 8 to day 30
  Evaluation of the game by healthcare professionals. Questionnaire of 6 questions of 7-level ordinal scale of answer, the higher the score, the more positive the appreciation ; 0 is the worst feeling and 100 the best.

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Fauroux, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No